CLINICAL TRIAL: NCT02615574
Title: A Phase 2 Study of Type-1 Polarized Dendritic Cell (αDC1) Vaccine in Combination With Tumor-Selective Chemokine Modulation (Interferon-α2b, Rintatolimod, and Celecoxib) in Subjects With Chemo-Refractory Metastatic Colorectal Cancer
Brief Title: A Study of Type-1 Polarized Dendritic Cell (αDC1) Vaccine in Combination With Tumor-Selective Chemokine Modulation (Interferon-α2b, Rintatolimod, and Celecoxib) in Subjects With Chemo-Refractory Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to inadequate supply of drug
Sponsor: Pawel Kalinski (Other)
Responsible Party: Sponsor-Investigator, Pawel Kalinski, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-023
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib; Introns; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- αDC1 vaccine + CKM (Experimental): all subjects enrolled in study
  Interventions: Biological: αDC1 vaccine; Drug: CKM

INTERVENTIONS:
Biological: αDC1 vaccine — Subjects will receive one cycle of CKM alone followed by three cycles of vaccine + CKM.
  Other Names: alpha-type-1-polarized dendritic cell vaccine
Drug: CKM — Subjects will receive one cycle of CKM alone followed by three cycles of vaccine + CKM.
  Other Names: celecoxib (Celebrex®); Interferon-α2b (IFN); rintatolimod (Ampligen®)

SUMMARY:
The investigators hypothesize that the treatment of metastatic colorectal cancer (mCRC) patients with the combination of alpha-type-1-polarized dendritic cell (αDC1) vaccines and tumor-selective chemokine modulation (CKM) will promote the infiltration of vaccination-induced CD8+ CTLs to tumor lesions and subsequently tumor regression with improved patient survival.

DETAILED DESCRIPTION:
Metastatic colorectal cancer is a major health concern in the United States, and the second leading cause of death due to cancer. The purpose of this trial is to see if the combination of the study vaccine and drugs in patients with this disease can prevent the growth of cancer and prevent new tumors from growing. The study drugs are a combination of celecoxib (Celebrex®), Interferon-α2b (IFN), and rintatolimod (Ampligen®), or CKM.

ELIGIBILITY:
Inclusion Criteria:

* Be age equal to 18 years or older.
* Be able to understand and be willing to sign a written informed consent document.
* Be HLA-A2 positive.
* Have mCRC that has been treated with currently approved standard therapies, including fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if KRAS wild type, an anti-EGFR therapy.
* Have at least 1 of the tumor sites that must be amenable to core needle biopsy and this may not be the site of disease used to measure antitumor response.
* Have measurable disease based on irRC.
* Have a performance status of ECOG 0 or 1.Have normal organ and marrow function as defined below:

  * Platelet ≥ 75,000/µL
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute Neutrophil Count (ANC) ≥ 1500/µL
  * Creatinine < 1.5 x institutional upper limit of normal (ULN) OR creatinine clearance (CrCl) ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels greater than 1.5 x ULN
  * Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) ≤ 2.5 x institutional upper limit of normal (ULN) OR

    ≤ 5 x ULN for subjects with liver metastases
  * Serum amylase and lipase within normal limits.

Exclusion Criteria:

* Is currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease or history of transplantation.
* Is a woman of child bearing potential (WOCBP) who are pregnant or nursing.
* Has a history of cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent. Subjects with a New York Heart Association classification of III or IV.
* Has a history of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years. Subjects with ulceration, bleeding or perforation in the lower bowel are not excluded.
* Has prior allergic reaction or hypersensitivity to celecoxib, or NSAIDs.
* Has an active infection requiring systemic therapy.
* Has significant ascites or pleural effusion requiring drainage for symptom relief.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C infection.
* Has history of asthma, or other allergic-type reactions after taking aspirin or other NSAIDs.
* Has known serious hypersensitivity reactions to peg-interferon alfa-2b or interferon alfa-2b.
* Has autoimmune hepatitis.
* Has hepatic decompensation (Child-Pugh score > 6; = class B and C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 36 months

SECONDARY OUTCOMES:
immune-related Overall Response Rate (irORR) | up to 36 months
immune-related Progression-Free Survival (irPFS) | up to 36 months

OTHER OUTCOMES:
Changes of CD8+ tumor infiltrating lymphocytes (CTLs) | up to 4 months
  Changes in CD8+ CTLs in paired tumor tissues collected at pre- and post-treatment.
Changes of tumor microenvironment | up to 4 months
  Changes of tumor microenvironment in paired tumor tissues collected at pre- and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James J Lee, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States